CLINICAL TRIAL: NCT02613156
Title: Efficacy Analysis of Complete Laparoscopic Resection of Recurrent Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongguo Zhou, Dr., Sun Yat-sen University
Other Study IDs: B20140001
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Recurrent Hepatocellular Carcinoma
Keywords: laparoscopic; hepatocellular carcinoma; recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- laparoscopic group: patients in the laparoscopic group underwent laparoscopic resection of recurrent HCC
  Interventions: Procedure: laparoscopic resection
- control group: patients in the control group underwent conventional open surgery

INTERVENTIONS:
Procedure: laparoscopic resection — The surgical instruments used for the laparoscopic group included conventional laparoscopic instruments (three 5 mm trocars, two 10 mm trocars, and two damage-free laparoscopic clamps), the STORZ high-resolution laparoscopic operating system (Germany), the GEN300 ultrasonic scalpel system (Johnson & Johnson, USA), a laparoscopic linear cutter stapler (Johnson & Johnson, USA), a laparoscopic ultrasound device, LigaSure, bipolar coagulation, titanium laparoscopic clips, and absorbable hemostatic gauze.
  Groups: laparoscopic group

SUMMARY:
This study is aiming to evaluate the clinical efficacy of complete laparoscopic resection of recurrent hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
The investigators conducted a prospective study of 64 patients who were diagnosed with recurrent HCC and underwent surgical resection at the Sun Yat-sen University Cancer Center from June 2014 to November 2014; 31 patients were enrolled in the laparoscopic group and underwent complete laparoscopic resection of HCC, and 33 patients were enrolled in the control group and underwent open surgical resection. The operation time, intraoperative blood loss, shortest distance between the tumor edge and normal liver tissue, postoperative pain scores, postoperative time until the patient could walk, postoperative time until the patient could pass gas, hospital stay, and inpatient costs were compared between the two groups. The patients were followed up for one year after surgery, and the relapse-free survival was compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. recurrent HCC after open surgery
2. recurrent HCC located in any part of the left lateral lobe or the diaphragm side of the right lobe and near the surface of the liver, which resulted in an easier operation
3. no significant surgical contraindications
4. no major vessel or bile duct tumor invasion and metastasis
5. grade A or B liver function or grade C liver function that recovered to grade A after liver-protective treatment;
6. the patient and his/her family was willing to undergo laparoscopic resection.

Exclusion Criteria:

1. major vessel or bile duct tumor invasion
2. recurrent HCC located in the right liver parenchyma and near secondary vessels and bile ducts, resulting in a difficult operation
3. grade C liver function
4. significant surgical contraindications
5. the patient and his/her family declined laparoscopic hepatectomy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were diagnosed with recurrent HCC and underwent surgical resection at the Sun Yat-sen University Cancer Center from June 2014 to November 2014
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Perioperative complications | within the first 30 days
  The operation time, intraoperative blood loss, shortest distance between the tumor edge and normal liver tissue, postoperative pain scores, postoperative time until the patient could walk, postoperative time until the patient could pass gas, hospital stay, and inpatient costs were compared between the two groups.

SECONDARY OUTCOMES:
relapse-free survival | 1 year after surgery
  The patients were followed up for one year after surgery, and the relapse-free survival was compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Li Xu, Study Director — Sun Yat-sen University